CLINICAL TRIAL: NCT06267924
Title: SENSE-VM: Safety and Effectiveness of a Novel Medical Device for Symptom Ease in Vestibular Migraines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otolith Labs (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Olith10703
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Vestibular Migraine; Migraine Associated Vertigo

STUDY DESIGN:
Intervention Model Description: The proposed clinical trial for the study device will be a randomized, sham-controlled, double-blind study with two-parallel arms (active/sham device).
Who Masked: Participant, Investigator
Masking Description: Clinical Research Coordinators, Clinical Trial Manager, Clinical Team Lead, and other members of the Sponsor organization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 1. Moderate or Worse (MoW) Arm (Experimental): Participants will be randomized to use the Otoband as instructed by clinical coordinator per study protocol. These participants will receive the experimental treatment device.
  Interventions: Device: Otoband Experimental
- 2. Moderate or Worse (MoW) Arm (Sham Comparator): Participants will be randomized to use the Otoband as instructed by clinical coordinator per study protocol. These participants will receive the sham device.
  Interventions: Device: Otoband Sham

INTERVENTIONS:
Device: Otoband Experimental — Participants will be randomly assigned to use the Otoband Experimental device to determine effectiveness in providing temporary relief to symptoms of vertigo.
  Arms: 1. Moderate or Worse (MoW) Arm
Device: Otoband Sham — Participants will be randomly assigned to use the Otoband Sham device to determine effectiveness in providing temporary relief to symptoms of vertigo.
  Arms: 2. Moderate or Worse (MoW) Arm

SUMMARY:
The goal of this virtual clinical trial is to compare the effectiveness of two study devices in providing temporary relief to adults aged 18-75 who suffer from symptoms of chronic Vestibular Migraines (VM), also known as Migraine Associated Vertigo.

Participants will be:

* Enrolled up to 50 days; enrollment, 14 days in Baseline Phase (no device), 7 days in Transition Phase, 28 days in Treatment Phase (study device)
* Randomized and stratified into groups based on the referring clinic to be assigned one study device
* Asked to use the study device as instructed by the study coordinator
* Asked to submit daily diaries reporting their symptoms and use of device, and to participate in tele-health visits with study coordinators
* Asked to provide their vertigo diagnosis from their physician
* Compensated for their participation

Researchers will compare the randomized groups to determine which group responds better to which device.

DETAILED DESCRIPTION:
This study is a decentralized clinical trial. This study uses technology and virtual meetings to communicate with study participants and collect study data. This study seeks to enroll until 200 participants have completed the study per protocol.

Study participants that meet all of the inclusion, none of the exclusion criteria, and sign the informed consent form will be enrolled in the study. Participants will complete a one day enrollment meeting and a 14 day Baseline Phase.

If a participant is eligible to remain in the study for the Treatment Phase at day 15, they will be randomized within their assigned group at a 1:1 ratio to an Active arm or Sham arm to begin the Treatment Phase of the study. Participants will be sent a study device to use when they have a vertigo episode.

Participants that enroll in the study are expected to participate up to 50 days with virtual meetings at the approximate intervals:

Day 5, Day 15, Day 22, Day 25, Day 35, and Day 51

Participants will be required to complete the DHI (Dizziness Handicap Inventory), VM-PATHI (Vestibular Migraine Patient Assessment Tool and Handicap Inventory), General Vertigo History, Global Impression of Change, "Most Bothersome Symptom", Relief from "Most Bothersome Symptom", and Net promoter score questionnaires.

Otolith Labs received Therapeutic Breakthrough Device designation by the FDA in May 2021.

ELIGIBILITY:
Inclusion Criteria:

To be eligible to participate in this study, an individual must meet all the following criteria:

- Diagnosed as having Vestibular Migraine (VM) (aka Migraine Associated Vertigo) The participant's diagnosis must be provided by a physician, Board certified in Otolaryngology or Neurology, from one of the study's approved clinics.

Diagnosis for VM must follow Bárány Society's "International Classification of Vestibular Disorders", which contains the Society's consensus diagnostic criteria for VM [Lempert 2022, sect. 3].

* Male or female subjects, age 18 to 75 years old inclusive on day of enrollment
* Residing in the United States
* Vestibular migraines that have been recurrent for at least 90 days
* Score from 36 to 90 inclusive on the Dizziness Handicap Inventory (DHI) (corresponding to moderate to severe vertigo)
* A smartphone, computer or tablet and access to internet to complete study procedures and study meetings
* Willing and able to comply with study procedures
* Willingness to use Venmo or Paypal for study stipend

Exclusion Criteria:

* Females who are pregnant or trying to become pregnant
* Enrolled in previous Otolith Lab-sponsored clinical trial
* Currently taking part in another interventional trial
* Surgery to the skull base within the last 6 months or plans for surgery to the skull during enrollment period
* Skull or neck implants
* History of vitreous detachment in the last 90 days
* Superior canal dehiscence or otic capsule dehiscence
* Diagnosed hyperacusis
* Planning to start vestibular rehabilitation therapy during the study
* History of cerebrovascular disorders
* Posterior fossa tumors, vestibular schwannoma
* Cerebellar degeneration (progressive worsening of neurons behind the brain stem)
* Initiation of calcitonin gene-related peptide inhibitor treatment within 4 weeks prior to beginning of trial
* Cognitive impairment or inability to follow study procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-01-08 (Actual)

PRIMARY OUTCOMES:
DHI Change in Scores | Day 23 - Day 51
  Reduction in final "Dizziness Handicap Inventory" (DHI) score by at least 12 points, compared to transition DHI score

SECONDARY OUTCOMES:
Number of related adverse events | Day 23 - Day 51
  Assessment of any adverse events related to device usage
Change in number of vestibular migraine episodes weekly | Day 1 - Day 51
  Assessment of the number of vestibular migraine episodes each week
Global Impression of Change (severity of episodes) | Day 51
  Assessment of the results of Global Impression of Change questionnaire and impacts on the severity of episodes
DHI change from transition to end of study | Day 23 - Day 51
  Assessment of overall changes in DHI score from transition time point to the end of the study
Device responder rate | Day 23 - Day 51
  Assessment of the responder rate of the study arms and their device usage

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Principal Investigator — Otolith Labs
Locations (1):
- Otolith Labs, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be made available to other researchers in an aggregate fashion upon publication of this study.